CLINICAL TRIAL: NCT06459219
Title: Factors Determining Tolerance to Nasal Allergen Exposure With Advanced Age in a Subset of Birch Pollen Allergic Subjects
Acronym: AllergyAge
Status: Not yet recruiting | Type: Observational
Sponsor: Sven Schneider, MD (Other)
Responsible Party: Sponsor-Investigator, Sven Schneider, MD, MD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: AllergyAge
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Allergic Rhinitis; Allergic Conjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Nasal secretions, nasal biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Ongoing (symptoms min 3 years): Ongoing intermittent allergic rhinoconjunctivitis to birch pollen with moderate to severe symptoms according to ARIA guidelines for at least 10 years Positive Skin prick test (SPT) to birch pollen and/or Bet v 1-specific IgE ≥0.35kUA/L as measured by ImmunoCAP
  ≥60 y
- Previous (no symptoms past 3 years): History of intermittent allergic rhinoconjunctivitis to birch pollen ongoing with moderate to severe symptoms according ARIA guidelines26 for at least ten years (verified by at least one medical record including SPT results), but no symptoms for at least the three past consecutive seasons Positive or negative SPT to birch pollen and Bet v 1-specific IgE ≤ or ≥0.35kUA/L as measured by ImmunoCAP
  ≥60 y
- No (never symptoms): No history of and no ongoing allergic rhinoconjunctivitis to birch pollen Negative SPT to birch pollen and Bet v 1-specific IgE ≤ 0.35kUA/L
  ≥60 y

SUMMARY:
Nasal allergen study in patients aged 60+ with or without current respiratory allergy

DETAILED DESCRIPTION:
Allergic rhinoconjunctivitis (AR) represents a major health burden affecting an estimated 1.4 billion people globally. It is characterized by inflammation of the nasal mucosa and conjunctiva in response to exposure to airborne allergens (e.g. pollen, dust mites). Interestingly, with advanced age, prevalence of AR decreases suggesting that a subset of allergic patients is able to develop tolerance towards allergens resulting in absence of symptoms. Understanding this mechanism governing natural tolerance development in the context of allergy is critical for the development of new therapeutic approaches and thus the aim of the proposed study. To address this question, the investigators plan to conduct a nasal allergen challenge study in patients aged 60+ who (1) are currently suffering from birch pollen allergy, (2) have a history of birch pollen allergy but absence of symptoms for at least three seasons and (3) never suffered from birch pollen allergy. After signing informed consent and fulfilling selection criteria, 38 patients per group will be intranasally challenged with birch pollen extract outside of the birch pollen season (October) and followed closely for up to 10 weeks to assess clinical parameters, cytokines, allergen-specific Immunoglobulin (Ig) levels as well as inflammatory cell subsets under controlled pollen exposure. In summary, this study will yield important information on the mechanisms underlying natural tolerance development in respiratory allergy with advanced age.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria Age ≥ 60 years Willingness to participate in the study and to follow the protocol Written informed consent Standard healthcare insurance Subjects should be available during the entire study period
* Patient group specific inclusion criteria (n=38 per group):

  1. Group 1 (current allergy):

     Ongoing intermittent allergic rhinoconjunctivitis to birch pollen with moderate to severe symptoms according to ARIA guidelines for at least 10 years Positive Skin prick test (SPT) to birch pollen and/or Bet v 1-specific IgE ≥0.35kUA/L as measured by ImmunoCAP
  2. Group 2 (former allergy):

     History of intermittent allergic rhinoconjunctivitis to birch pollen ongoing with moderate to severe symptoms according ARIA guidelines for at least ten years (verified by at least one medical record including SPT results), but no symptoms for at least the three past consecutive seasons Positive or negative SPT to birch pollen and Bet v 1-specific IgE ≤ or ≥0.35kUA/L as measured by ImmunoCAP
  3. Group 3 (never allergy):

No history of and no ongoing allergic rhinoconjunctivitis to birch pollen Negative SPT to birch pollen and Bet v 1-specific IgE ≤ 0.35kUA/

Exclusion Criteria:

* - Evidence of acute, chronic, malignant or general diseases-assessed by asking the patient
* A History of anaphylaxis
* Utilization of leukotriene modifiers or long-acting antihistamines
* Chronic or intermittent use of oral, inhaled, intramuscular or intravenous corticosteroids
* Nasal polyps, history of chronic sinusitis or considerable deviation of the nasal septum
* Rhinitis secondary to other causes
* Contra-indications to skin prick testing, for example, skin irritation in the test area and urticaria facticia
* Cardiovascular diseases requiring treatment with anti-hypertensive medication or beta-blockers
* Known clotting disorders
* Chronic use of additional medications that would affect assessment and the results of the study (e.g., tricyclic antidepressants that block both H1 and H2 receptors)
* Pregnant or breastfeeding females
* Actual disability that would influence subject's ability to participate in the study
* History of mental illness, intellectual deficiency, drug or alcohol abuse
* Active asthma requiring treatment
* Allergen immunotherapy within the last 5 years to any allergen
* Current and former smokers who stopped smoking <1 year ago

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 60 years with or without current or former allergy
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Nasal IgG4 | 5 weeks
  To demonstrate that Bet v 1-specific nasal IgG4 responses 5 weeks after controlled nasal birch pollen provocation are significantly higher in subjects aged ≥60y without ongoing respiratory allergic symptoms with a history of allergy (group1) as compared to age-matched subjects currently suffering from allergic rhinoconjunctivitis (group 2).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided